CLINICAL TRIAL: NCT04948593
Title: The Risks of Percutaneous Native Kidney Biopsy in Italy in the Third Millennium: a Prospective Cohort Study
Brief Title: The Risks of Percutaneous Native Kidney Biopsy in Italy: a Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Simeone Andrulli, MD (Other)
Responsible Party: Sponsor-Investigator, Simeone Andrulli, MD, Simeone Andrulli, MD, A. Manzoni Hospital
Organization: A. Manzoni Hospital (Other)
Other Study IDs: KidneyBiopsyRisk in Italy
Record Dates: First submitted 2021-06-07; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Native kidney biopsy

SUMMARY:
The estimates risks and benefits of the percutaneous kidney biopsy have been reported mainly from retrospective studies. So far no prospective multicentre studies has been designed to identify rates of biopsy related complications. The aim of this prospective multicentre study was to evaluate safety and complication events related to biopsies on native kidney in Italy.

DETAILED DESCRIPTION:
Kidney biopsies performed in 54 italian nephrology centres from 2012 to 2020 were included.

Primary outcome of the study was any major complication, such as haemoglobin decrease more than 2 g/dL, macroematuria, gross ematoma, blood transfusion, artero-venous fistula, invasive intervention, pain, symptomatic hypotension, and/or rapid serum creatinine increase.

Centre and individual patient risk predictors were analysed using multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult or pediatric patients with a kidney disease
* informed Consent

Exclusion Criteria:

* patient with a transplanted kidney

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data collection of native kidney biopsies was centralized and takes place via Web by means of an ad hoc web-database linked to the National Italian Renal Biopsy Registry (http://www.irrb.net/). As this is an observational study, we collect information already available and typical of usual clinical practice. There are no particular requested exams.
Sampling Method: Non-Probability Sample
Enrollment: 5304 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Any major post-biopsy complication event | one week follow-up after native kidney biopsy
  The cecked of major post-biopsy complication events were clinically relevant hematomas, macrohematuria, decrease of haemoglobin levels after 24 hours > 2 g /dL, the need for blood transfusion, a large and persistent AV fistula, a post-biopsy anuria, an increase in serum creatinine greater than 50% in the week following biopsy, the need for invasive post-biopsy procedure related to the procedure including nephrectomy, the death related to biopsy

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (18):
  - San Giovanni di Dio Hospital, Agrigento
  - Giovanni XXIII pediatric Hospital, Bari
  - Policlinico Hospital, Bari
  - S. Orsola Hospital, Bologna
  - Cannizzaro Hospital, Catania
  - S. Camillo Hospital, Chieti
  - Santa Croce Hospital, Cuneo
  - Maria SS. Addolorata Hospital, Eboli
  - University Hospital, Foggia
  - Policlinico Hospital, Messina
  - Cervello Hospital, Palermo
  - Riuniti Hospital, Parma
  - Ospedali Riuniti Marche Nord Hospital, Pesaro
  - Cisanello Hospital, Pisa
  - Umberto 1° Hospital, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Sollievo Sofferenza Hospital, San Giovanni Rotondo
  - Belcolle Hospital, Viterbo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Italian Registry Renal Biopsy — http://www.irrb.net/